CLINICAL TRIAL: NCT03298620
Title: Effect of Electric Toothbrush on Oral Hygiene in Nursing Home Residents- a Randomized Clinical Trial
Brief Title: Electric and Manual Toothbrushes in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Tiril Willumsen, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC-2011/915-5
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Oral Health
Keywords: nursing home; gerodontology; oral hygiene

STUDY DESIGN:
Intervention Model Description: Randomized Clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: A dental team (dentist and dental hygienist) assessed the outcome measure at baseline and after the two months RCT trial. A neutral dentist implements the intervention after baseline registration. Toothbrushes used in the intervention period is hidden to the dental team during assessments at the end of the RCT period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Electric toothbrush
  Interventions: Other: Electric toothbrush
- Control (Active Comparator): New standard manual toothbrush
  Interventions: Other: Control

INTERVENTIONS:
Other: Electric toothbrush
  Arms: Intervention
Other: Control — Manual toothbrush
  Arms: Control

SUMMARY:
Effect of electric toothbrush on oral hygiene in nursing home residents tested I randomized clinical trial for 2 months and followed up 12 months after baseline

DETAILED DESCRIPTION:
Patients in nursing homes often have many natural teeth with exposed root surfaces, bifurcations, a complexity of dental restorations like partial prostheses, bridges/crowns, fillings and implants. In addition they have a limited physical ability, like reduced muscular strength, rigidness in the neck and spine. All these factors contribute to make it difficult, both for themselves and their nursing staff to maintain good oral hygiene.

Electrical toothbrushes have been proved effective in removal of dental plaque. There have also been reports from nursing homes that approves of electrical toothbrushes as a helpful aid among the nursing staff.

The present study examine if the overall oral hygiene actually improves with the use of electric toothbrush.

Material and method: The study is a randomized clinical trial (RCT) that includes patients from nursing homes in Oslo. The recording dentist is blind to the type of tooth brush Inclusion criteria.

* Patients living in nursing home in Oslo
* Provide written informed consent prior to enrolment (from relatives when patients were assessed by physician to be without ability to give written consent.

Participants in the experimental group use an electrical toothbrush. Participants in the control group use a standard manual toothbrush.

Registration of oral hygiene and plaque score at baseline 0 and after 2 months intervention.

After the RCT trial the participants were free to choose toothbrush, electric or manual. The study includes a follow-up study 10 months after the end of the RCT trial.

The study is a part of the PhD programme for Katrine Gahre Fjeld Cand. Odont.

Supervisors:

Tiril Willumsen Dr Odont, The Dental Faculty, University of Oslo Hilde Eide Dr. Philos, Department of Nursing, Buskerud University College Morten Mowe Dr med, The Medical Faculty, University of Oslo

ELIGIBILITY:
Inclusion Criteria:

* Patients living in nursing home in Oslo
* Provide written informed consent prior to enrolment (from relatives when patients were assessed by physician to be without ability to give written consent.

Exclusion Criteria:

* Patients too weak to be examined
* Patients With life expectancy less then one year

Ages: 70 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 233 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Change in dental plaque score by use of the Oral Hygiene Index- simplified (OHI-S) | baseline, after 2 months, after 12 months
  OHI-S is measuring amount of dental plaque using 6 indicator teeth. Outcome measure: change in OHI-S

CONTACTS AND LOCATIONS:
Overall Officials: Tiril Willumsen, Principal Investigator — Institute of Clinical Odontology
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Background] Samson H, Strand GV, Haugejorden O. Change in oral health status among the institutionalized Norwegian elderly over a period of 16 years. Acta Odontol Scand. 2008;66(6):368-73. doi: 10.1080/00016350802378654. PMID 18792846
- [Background] Meurman JH, Hamalainen P. Oral health and morbidity--implications of oral infections on the elderly. Gerodontology. 2006 Mar;23(1):3-16. doi: 10.1111/j.1741-2358.2006.00102.x. PMID 16433636
- [Background] Hamalainen P, Meurman JH, Kauppinen M, Keskinen M. Oral infections as predictors of mortality. Gerodontology. 2005 Sep;22(3):151-7. doi: 10.1111/j.1741-2358.2005.00064.x. PMID 16163906
- [Background] Zuluaga DJ, Ferreira J, Montoya JA, Willumsen T. Oral health in institutionalised elderly people in Oslo, Norway and its relationship with dependence and cognitive impairment. Gerodontology. 2012 Jun;29(2):e420-6. doi: 10.1111/j.1741-2358.2011.00490.x. Epub 2011 May 12. PMID 21564272
- [Background] Henriksen BM, Ambjornsen E, Axell T. Dental caries among the elderly in Norway. Acta Odontol Scand. 2004 Apr;62(2):75-81. doi: 10.1080/00016350310008580. PMID 15198386
- [Background] Wolden H, Strand GV, Gjellestad A. Caregivers' perceptions of electric versus manual toothbrushes for the institutionalised elderly. Gerodontology. 2006 Jun;23(2):106-10. doi: 10.1111/j.1741-2358.2006.00114.x. PMID 16677184
- [Background] Forrest JL, Miller SA. Manual versus powered toothbrushes: a summary of the Cochrane Oral Health Group's Systematic Review. Part II. J Dent Hyg. 2004 Spring;78(2):349-54. PMID 15190692
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Background] Henriksen BM, Ambjornsen E, Axell TE. Evaluation of a mucosal-plaque index (MPS) designed to assess oral care in groups of elderly. Spec Care Dentist. 1999 Jul-Aug;19(4):154-7. doi: 10.1111/j.1754-4505.1999.tb01378.x. PMID 10765880
- [Background] Lindqvist L, Seleskog B, Wardh I, von Bultzingslowen I. Oral care perspectives of professionals in nursing homes for the elderly. Int J Dent Hyg. 2013 Nov;11(4):298-305. doi: 10.1111/idh.12016. Epub 2013 Feb 25. PMID 23433346
- [Background] Robinson PG, Damien Walmsley A, Heanue M, Deacon S, Deery C, Glenny AM, Worthington H, Shaw W. Quality of trials in a systematic review of powered toothbrushes: suggestions for future clinical trials. J Periodontol. 2006 Dec;77(12):1944-53. doi: 10.1902/jop.2006.050349. PMID 17209777
- [Background] Deery C, Heanue M, Deacon S, Robinson PG, Walmsley AD, Worthington H, Shaw W, Glenny AM. The effectiveness of manual versus powered toothbrushes for dental health: a systematic review. J Dent. 2004 Mar;32(3):197-211. doi: 10.1016/j.jdent.2003.11.006. PMID 15001285
- [Background] Robinson PG, Deacon SA, Deery C, Heanue M, Walmsley AD, Worthington HV, Glenny AM, Shaw WC. Manual versus powered toothbrushing for oral health. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD002281. doi: 10.1002/14651858.CD002281.pub2. PMID 15846633
- [Background] Hagman-Gustafsson ML, Holmen A, Stromberg E, Gabre P, Wardh I. Who cares for the oral health of dependent elderly and disabled persons living at home? A qualitative study of case managers' knowledge, attitudes and initiatives. Swed Dent J. 2008;32(2):95-104. PMID 18700337
- [Background] Stromberg E, Hagman-Gustafsson ML, Holmen A, Wardh I, Gabre P. Oral status, oral hygiene habits and caries risk factors in home-dwelling elderly dependent on moderate or substantial supportive care for daily living. Community Dent Oral Epidemiol. 2012 Jun;40(3):221-9. doi: 10.1111/j.1600-0528.2011.00653.x. Epub 2011 Nov 9. PMID 22070521
- [Background] Philip P, Rogers C, Kruger E, Tennant M. Caries experience of institutionalized elderly and its association with dementia and functional status. Int J Dent Hyg. 2012 May;10(2):122-7. doi: 10.1111/j.1601-5037.2011.00525.x. Epub 2011 Aug 5. PMID 21815998
- [Background] Arpin S. Oral hygiene in elderly people in hospitals and nursing homes. Evid Based Dent. 2009;10(2):46. doi: 10.1038/sj.ebd.6400649. PMID 19561578
- [Background] Willumsen T, Fjaera B, Eide H. Oral health-related quality of life in patients receiving home-care nursing: associations with aspects of dental status and xerostomia. Gerodontology. 2010 Dec;27(4):251-7. doi: 10.1111/j.1741-2358.2009.00344.x. PMID 19780842
- [Background] Haumschild MS, Haumschild RJ. The importance of oral health in long-term care. J Am Med Dir Assoc. 2009 Nov;10(9):667-71. doi: 10.1016/j.jamda.2009.01.002. Epub 2009 Jun 28. PMID 19883892
- [Background] Marsh PD. Contemporary perspective on plaque control. Br Dent J. 2012 Jun 22;212(12):601-6. doi: 10.1038/sj.bdj.2012.524. PMID 22722123